CLINICAL TRIAL: NCT04137393
Title: The Effect of Brushing With Salvadorapersica (Miswak) Sticks on Salivary Streptococcus Mutants and Plaque Level in Children: A Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heba sabbagh (Other)
Responsible Party: Sponsor-Investigator, Heba sabbagh, assistant professor, King Abdulaziz University
Organization: King Abdulaziz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 006-16
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salvadora persica (Experimental): brush teeth with Salvadora persica "Miswak"
  Interventions: Combination Product: brushing
- tooth brush (Active Comparator): brush with fluoridated tooth paste
  Interventions: Combination Product: brushing

INTERVENTIONS:
Combination Product: brushing — mechanical and chemical plaque removal

SUMMARY:
Objectives:

to evaluate the effect of brushing with Salvadora persica (Miswak) on streptococcus mutants compared to brushing with fluoridated tooth paste (FTP) in children.

Methods:

A total of 94 healthy children (8 years old) from an elementary governmental school in Jeddah, Saudi Arabia were grouped to Miswak and FTP groups. They were assessed for their salivary level of mutans streptococci species, and lactobacillus at the baseline and three weeks after brushing. Caries level using DMFT/dmft, and plaque amount using Greene Vermillion simplified oral hygiene index were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* age from 8 to 9
* parents signed the consent form they attended morning session for brushing

Exclusion Criteria:

* medical compromised children
* parents did not sign the consent form Did not attend morning session

Ages: 8 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
green and vermillion | 4 months
  plaque level

REFERENCES:
- [Derived] Sabbagh HJ, AlGhamdi KS, Mujalled HT, Bagher SM. The effect of brushing with Salvadora persica (miswak) sticks on salivary Streptococcus mutans and plaque levels in children: a clinical trial. BMC Complement Med Ther. 2020 Feb 13;20(1):53. doi: 10.1186/s12906-020-2847-3. PMID 32054468